CLINICAL TRIAL: NCT07339371
Title: A Prospective Cohort Study on Comprehensive Care of Sleep Disordered Breathing (Care-SDB Study)
Brief Title: Comprehensive Care of Sleep Disordered Breathing
Acronym: Care-SDB
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Second Xiangya Hospital of Central South University (Other); Peking University Hospital of Stomatology (Other); Shantou University Medical College (Other); Shanghai Institute of Hypertension (Other); First Affiliated Hospital of Fujian Medical University (Other); Beijing Tiantan Hospital (Other); Beijing Jishuitan Hospital (Other); Beijing Friendship Hospital (Other); West China Hospital (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Shao-Ping Nie, Professor of Medicine, Beijing Anzhen Hospital
Other Study IDs: KS2025041
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sleep Disordered Breathing (SDB)
Keywords: Comprehensive Care; Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SDB Comprehensive Management Cohort: This is a multi-center, prospective, observational registration cohort of 11,100 adult patients (age ≥ 18). All participants must have completed sleep breathing monitoring within one month prior to enrollment. The cohort aims to establish a clinical database and biobank to explore SDB-related biomarkers and pathogenesis. Participants receive comprehensive clinical management, including potential treatments for SDB, such as continuous positive airway pressure (CPAP), oral appliances, surgery, or lifestyle interventions. Data on clinical baselines, sleep monitoring, laboratory tests, and imaging will be collected. Follow-up will be conducted for up to 5 years (at baseline, 3 months, 1 year, and annually thereafter) to evaluate clinical outcomes, including all-cause mortality and cardiovascular events.
  Interventions: Other: Clinical Management for SDB

INTERVENTIONS:
Other: Clinical Management for SDB — Participants receive standard clinical care and management for sleep-disordered breathing according to established clinical guidelines. This may include, but is not limited to, CPAP therapy, lifestyle modifications, oral appliances, or other medical interventions as determined by the treating physician.

SUMMARY:
The Comprehensive Care of Sleep Disordered Breathing study (Care-SDB) is a prospective, multi-center, registry-based cohort study designed to investigate the integrated management of sleep-disordered breathing (SDB). The investigators aim to establish a nationwide SDB cohort and biobank to identify prognostic biomarkers, explore pathogenic mechanisms, and evaluate optimal treatment models. A total of 11,100 adult patients with recent sleep monitoring will be enrolled and followed longitudinally for up to 5 years. Data collection, including clinical outcomes and major adverse events, will be managed via a unified Electronic Data Capture platform. The results from Care-SDB are expected to provide critical evidence-based guidance for the risk stratification, standardized intervention, and personalized management of patients with sleep-disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients who have completed sleep breathing monitoring within 1 month prior to enrollment.
* Capable of providing signed informed consent.

Exclusion Criteria:

* Estimated life expectancy of less than 3 months.
* Refusal to participate in the study.
* Inability to cooperate with baseline data collection or follow-up evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients presenting to the outpatient or inpatient departments of participating clinical centers across China who have completed or are scheduled for sleep breathing monitoring for suspected or confirmed SDB.
Sampling Method: Non-Probability Sample
Enrollment: 11100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 3 and 12 months after enrollment, then annually thereafter, with a maximum follow-up duration of 5 years

SECONDARY OUTCOMES:
All-cause hospitalization | Up to 5 years.
Comorbidity-related Adverse Events | Up to 5 years.
  Major adverse cardiovascular and cerebrovascular events (MACCE, a composite endpoint including cardiac mortality, non-fatal myocardial infarction, non-fatal stroke, ischemia-driven revascularization and readmission due to angina), the individual endpoints included in MACCE.
  Occurrence and recurrence of arrhythmias such as atrial fibrillation. Respiratory-related adverse events (chronic obstructive pulmonary disease exacerbation, asthma attacks, progression of interstitial lung disease, and pulmonary embolism, etc).
  Metabolism-related adverse events (diabetes, diabetic complications, non-alcoholic fatty liver disease, etc).
  Psychology-related adverse events (anxiety and depression, cognitive impairment, Alzheimer's disease, Parkinson's disease, epilepsy, etc).
  Chronic kidney disease-related adverse events (progression of renal function to end-stage renal disease, significant decline in estimated glomerular filtration rate, etc) Tumor occurrence and progression.
Change from Baseline in Sleep-Disordered Breathing Parameters | Baseline and up to 5 years.
  Evaluation of changes in parameters such as Apnea-Hypopnea Index (AHI) and Oxygen Desaturation Index (ODI) through repeated sleep breathing monitoring.
Change in Daytime Sleepiness assessed by Epworth Sleepiness Scale (ESS) | Baseline and up to 5 years.
  The ESS is a self-administered questionnaire with 8 questions. Each item is scored from 0 to 3, with a total score range of 0 to 24. Higher scores indicate increased daytime sleepiness, representing a worse outcome.
Quality of Life assessed by 36-Item Short Form Survey (SF-36) | Baseline and up to 5 years.
  The SF-36 Scale consists of eight scaled scores. Each scale is directly transformed into a 0-100 scale. Possible scores range from 0 to 100, where higher scores represent better health status or less disability, indicating a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China